CLINICAL TRIAL: NCT02979704
Title: Randomized. Open Label Trial of Comparison Between Rosuvastatin and Atorvastatin on Oxidative Stress, Inflammatory and Thrombogenic Biomarkers in Patients With Hyperlipidemia
Brief Title: A Comparative Study of Rosuvastatin and Atorvastatin in Patients With Hyperlipidemia
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Samia Haque Tonu, Dr. and MD resident, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: No.BSMMU/2016/8307
Record Dates: First submitted 2016-08-31; First posted 2016-12-02 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-08

CONDITIONS: Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias | interventions — Rosuvastatin Calcium; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rosuvastatin (Active Comparator): Intervention: Tablet Rosuvastatin (5-10) mg orally once daily dose for 08 weeks.
  Interventions: Drug: Rosuvastatin
- Atorvastatin (Active Comparator): Intervention: Tablet Atorvastatin (10-20) mg orally once daily dose for 08 weeks
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Rosuvastatin — 45 patients will be treated with rosuvastatin at a dose of (5-10) mg orally once daily dose for 08 weeks
  Other Names: Rocovas
  Arms: Rosuvastatin
Drug: Atorvastatin — 45 patients will be treated with atorvastatin at a dose of (10-20) mg orally once daily dose for 08 weeks
  Other Names: Tiginor
  Arms: Atorvastatin

SUMMARY:
This study will be conducted to assess the status of oxidative stress inflammation and thrombogenesis in patients with hyperlipidemia and to compare the antioxidative, anti-inflammatory and antithrombogenic effects of rosuvastatin and atorvastatin.

DETAILED DESCRIPTION:
Hyperlipidemia is the major risk factor for development of atherosclerosis which ultimately leads to cardiovascular disease (CVD), an important cause of mortality and morbidity worldwide. Atherosclerosis was previously considered as a lipid storage disease but now growing evidence indicates that increased oxidative stress, vascular inflammation and platelet activation play an important role in the initiation and progression of atherosclerosis. Among the hypolipidemic drugs, statins, 3-hydroxyl-3-methylglutaryl coenzyme A (HMG-CoA) reductase inhibitors, have proved to be very much effective. Therefore, statins are the most widely used hypolipidemic agents. Evidence shows that besides hypolipidemic action statins possess antioxidative, anti-inflammatory and antithrombogenic effects known as pleiotropic action which might play an important role in attenuating the atherosclerotic process. However, pleiotropic effect varies with different members of statins.

The present prospective interventional study would be conducted in the Department of Pharmacology, Department of Cardiology and Internal Medicine, BSMMU from March 2016 to August 2017. Total 90 cases will be selected according to inclusion and exclusion criteria. The cases will be subdivided into 2 groups: group A and B. Group A consisting of 45 patients who will receive rosuvastatin (5-10) mg orally once daily and Group B consisting of 45 patients who will receive atorvastatin (10-20) mg orally once daily for 08 weeks. Patient's blood sample will be collected to measure baseline lipid profile, malondialdehyde (MDA), erythrocytic glutathione (GSH), high sensitive C-reactive protein (hs-CRP), prothrombin time (PT), platelet count. After obtaining baseline data patients will be assigned to the respective group. Parameters of baseline will again be evaluated after 08 weeks of therapeutic intervention. Regularity of drug intake will be ensured over telephone, pill count, and from the patient's compliance sheet. Patient's data will be recorded in a predetermined data sheet. Patients will be informed about study, its merits and demerits in easy language and then informed consent will be taken.Therefore, the present study has been designed to compare the antioxidative, anti-inflammatory and antithrombogenic effects of rosuvastatin and atorvastatin in hyperlipidemic patients to establish the superiority of a particular statin, so that it will provide a better therapeutic option in order to prevent CVD related mortality and morbidity.

ELIGIBILITY:
Inclusion criteria:

* Age from (20-75) yrs, both male and female having LDL cholesterol: 160-190 mg/dl, triglyceride (TG): 200-499 mg/dl will be recruited in the study

Exclusion criteria:

* Patients age <25 years or >75 years
* Patients are on lipid lowering medications
* Patients taking omega-3 fatty acid or garlic
* Patients with history of hypersensitivity on any member of statin
* Patients taking anti-inflammatory medications (steroid or NSAIDS)
* Patients taking antioxidant vitamins (vitamin A, C, E)
* Patients with impaired renal function
* Patients with impaired liver function
* Pregnant women and nursing mother
* Patients having serious infections or terminal illness

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-06 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Establishment of superiority between rosuvastatin and atorvastatin on reduction of MDA in patients with hyperlipidemia | [0 weeks (baseline), 8 weeks (end)] [safety Issue: No]
  Reduction of oxidative stress will be measured by changes in level of MDA in µmol/L
Establishment of superiority between rosuvastatin and atorvastatin on reduction of inflammation in patients with hyperlipidemia | [0 weeks (baseline), 8 weeks (end)] [safety Issue: No]
  Reduction of inflammation will be measured by change in level of hs-CRP in mg/L
Establishment of superiority between rosuvastatin and atorvastatin on reduction platelet count in patients with hyperlipidemia | [0 weeks (baseline), 8 weeks (end)] [safety Issue: No]
  Reduction of thrombogenesis will be measured by changes in level of platelet count in per L of blood
Establishment of superiority between rosuvastatin and atorvastatin on increase prothrombin time in patients with hyperlipidemia | [0 weeks (baseline), 8 weeks (end)] [safety Issue: No]
  Reduction of thrombogenesis will be measured by changes in level of prothrombin time in per sec
Establishment of superiority between rosuvastatin and atorvastatin on increase level of erythrocytic GSH in patients with hyperlipidemia | [0 weeks (baseline), 8 weeks (end)] [safety Issue: No]
  Reduction of oxidative stress will be measured by changes in level of erythrocytic GSH in mg/gm of Hb

CONTACTS AND LOCATIONS:
Overall Officials: Samia Tonu, MBBS, Principal Investigator — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (1):
- BSMMU, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No